CLINICAL TRIAL: NCT05724472
Title: A Phase 1, Single-blind, Placebo-controlled, Dose-escalation Clinical Trial to Evaluate the Safety and Immunogenicity of rVSVΔG-SEBOV-GP Vaccine at 3 Dose Levels in Adults in Good General Health
Brief Title: Evaluation of Safety and Immunogenicity of rVSVΔG-SEBOV-GP Vaccine in Adults With Good General Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IAVI C108
Record Dates: First submitted 2023-01-05; First posted 2023-02-13 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Ebola Sudan Virus Disease

STUDY DESIGN:
Intervention Model Description: This is a single-blind, placebo-controlled, dose-escalation clinical trial to evaluate the safety and immunogenicity of rVSVΔG-SEBOV-GP vaccine at 3 dose levels in adults in good general health.
Who Masked: Participant
Masking Description: It is a single blind study. The participant will be unaware of the intervention.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Group 1 (Experimental): rVSV∆G-SEBOV-GP Vaccine or Placebo Dosage 2 × 10^6 pfu intramuscularly Day 1
  Interventions: Drug: rVSV∆G-SEBOV-GP Vaccine or Placebo
- Study Group 2 (Experimental): rVSV∆G-SEBOV-GP Vaccine or Placebo Dosage 2 × 10^7 pfu intramuscularly Day 1
  Interventions: Drug: rVSV∆G-SEBOV-GP Vaccine or Placebo
- Study Group 3 (Experimental): rVSV∆G-SEBOV-GP Vaccine or Placebo Dosage 2 × 10^8 pfu intramuscularly Day 1
  Interventions: Drug: rVSV∆G-SEBOV-GP Vaccine or Placebo

INTERVENTIONS:
Drug: rVSV∆G-SEBOV-GP Vaccine or Placebo — rVSV∆G-SEBOV-GP Vaccine or Placebo

SUMMARY:
A Phase 1, Single-blind, Placebo-controlled, Dose-escalation Clinical Trial to Evaluate the Safety and Immunogenicity of rVSVΔG-SEBOV-GP Vaccine at 3 Dose Levels in Adults in Good General Health

DETAILED DESCRIPTION:
The purpose of this study is to provide the needed safety and immunogenicity data to support rapid deployment of the SEBOV vaccine against an ongoing or future outbreak.

The intervention will be a single dose and will either be study vaccine named rVSVΔG-SEBOV-GP Vaccine, or placebo (a placebo is an inactive substance or other intervention that looks the same as and is given the same way as study vaccine or treatment being tested)

There are 3 group in this study, each group has different vaccine doses. Group 1 starts with the lowest dose of the study vaccine and each subsequent group Groups 2 and Group 3 gets a higher dose of the study vaccine.

Approximately 36 participants will be included in the study.

The participant will be unaware of the treatment given between placebo and study vaccine.

Participants will be screened up to 14 days before IP administration and will be followed for 6 months after IP administration. The anticipated study duration for each participant in Groups 1 through 3 is approximately 6.5 months from screening through last study visit.

ELIGIBILITY:
Inclusion:

* Good general health
* ≥18 years of age on the day of screening and are ≤50 years of age on the day of IP administration
* Adherence to the requirements of the protocol and the follow-up for the planned duration of the study
* Undergo HIV testing, risk reduction counseling, and receive HIV test results
* As applicable use male or female condoms for 1 month following IP administration
* Use an effective method of contraception from at least 2 weeks before and continue until 3 months following receipt of vaccine
* As applicable undergo urine pregnancy tests
* Forgo donation of blood or any other tissues throughout the course of the study

Exclusion:

* Any clinically relevant abnormality
* Any clinically significant acute or chronical medical condition
* Women who are pregnant or breastfeeding
* Bleeding disorder
* Infectious disease
* History of splenectomy
* Receipt of any vaccine within the previous 28 days or planned receipt within 28 days after vaccination with IP.
* Receipt of blood transfusion or blood-derived products within 3 months prior to screening
* Prior exposure to SEBOV or history of any hemorrhagic fever
* Prior receipt of any VSV-vectored vaccine
* Receipt of another IP within 3 months prior to enrollment or expected participation during this study.
* Prior receipt of another Sudan Ebola vaccine or receipt of polyclonal or monoclonal antibodies directed against Sudan Ebola in the past 6 months
* History of severe reactogenicity to vaccines or severe allergy to food or medications
* A history of malignancy in the past 5 years (prior to screening) or ongoing malignancy.
* Serious infections requiring antibiotic, antiviral, or antifungal therapy within 30 days prior to enrollment
* Body mass index (BMI) ≥35
* Current or planned occupational or household contact from screening through 3 months after vaccine administration with any immunocompromised individual

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of rVSVΔG-SEBOV-GP vaccine | 14 days
  Proportion of participants with Grade 3 or higher reactogenicity (ie, solicited AEs) during the 14 days after vaccine administration
To evaluate the safety and tolerability of rVSVΔG-SEBOV-GP vaccine | 14 days
  Proportion of participants with Grade 2 or higher vaccine-related unsolicited AEs, including safety laboratory parameters, within 14 days of vaccine administration
To evaluate the safety and tolerability of rVSVΔG-SEBOV-GP vaccine | 14 days
  Proportion of participants with Grade 2 or higher unsolicited AEs, including safety laboratory parameters, within 14 days of vaccine administration
To evaluate the safety and tolerability of rVSVΔG-SEBOV-GP vaccine | 14 days
  Proportion of participants with vaccine-related SAEs throughout the study period

SECONDARY OUTCOMES:
To determine SEBOV-GP-specific antibody responses induced by rVSVΔG-SEBOV-GP vaccine | 6.5 months
  Proportion of participants with binding antibody responses to SEBOV-GP
To determine SEBOV-GP-specific antibody responses induced by rVSVΔG-SEBOV-GP vaccine | 6.5 months
  Magnitude of binding antibody responses to SEBOV-GP
To determine SEBOV-GP-specific antibody responses induced by rVSVΔG-SEBOV-GP vaccine | 6.5 months
  Proportion of participants with neutralizing antibody responses against SEBOV
To determine SEBOV-GP-specific antibody responses induced by rVSVΔG-SEBOV-GP vaccine | 6.5 months
  Magnitude of neutralizing antibody responses against SEBOV

OTHER OUTCOMES:
To explore the characteristics of the immune responses induced by rVSV∆G-SEBOV-GP vaccine | 6.5 months
  Anti-GP IgG antibodies as measured in 'effector assays' such as ADCC
To explore the characteristics of the immune responses induced by rVSV∆G-SEBOV-GP vaccine | 6.5 months
  Anti-GP antibody epitope specificity
To explore the characteristics of the immune responses induced by rVSV∆G-SEBOV-GP vaccine | 6.5 months
  Anti-VSV-N antibodies
To explore the characteristics of the immune responses induced by rVSV∆G-SEBOV-GP vaccine | 6.5 months
  Additional exploratory immunological assessments may be conducted as warranted

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Benchmark Research, Austin, Texas
  - Clinical Trials of Texas, San Antonio, Texas

DOCUMENTS (1):
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT05724472/ICF_000.pdf